CLINICAL TRIAL: NCT06066736
Title: Risks Factors and Outcome of Recurrences in Patients With Ventilator-Associated Pneumonias (REVAP)
Acronym: REVAP
Status: Completed | Type: Observational
Sponsor: Société Française d'Anesthésie et de Réanimation (Other)
Responsible Party: Sponsor
Other Study IDs: REVAP / 2022-11
Record Dates: First submitted 2023-09-27; First posted 2023-10-04 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Ventilator-associated Pneumonia
MeSH Terms: conditions — Pneumonia, Ventilator-Associated | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with Ventilator-associated pneumonia: Patients having presented an episode of ventilator-associated pneumonia, undergoing invasive mechanical ventilation ≥ 48h
  Interventions: Other: observational

INTERVENTIONS:
Other: observational — No intervention, observational group

SUMMARY:
Ventilator-associated pneumonia (VAP) is a frequent and serious complication in the ICU, defined by the development of a lung infection in patients ventilated for more than 48 hours. The incidence rate of this condition exceeds 18 episodes per 1000 days of mechanical ventilation in Europe. This nosocomial infection is associated with the highest mortality, ranging from 24% to 76% depending on the series. Reducing the incidence of VAP remains a challenge for clinicians, as evidenced by the many recent recommendations that have led to "bundles" to prevent the onset of this complication. Despite this, these recommendations do not propose a strategy to prevent the recurrence of PAVM, a frequent entity with a reported incidence of 25-35% and a non-consensual definition that increases antibiotic consumption, duration of mechanical ventilation and length of stay in the ICU .

In fact, these recurrences can be linked to:

* Intrinsic patient risk factors (immunosuppression, severity of disease, major inflammatory response, reason for initial admission),
* Inappropriate initial antibiotic therapy (type, duration and dose administered),
* Characteristics specific to the pathogens encountered (virulence factors or resistance),
* Intercurrent complications during management of the initial pneumonia (ARDS, abscess, pleural empyema).

Given the frequency of these recurrences, and the persistent doubts about the role of terrain and pathogen characteristics in their genesis, it seems appropriate to look at risk factors that could help anticipate these events.

The aim of our study will be to identify the risk factors and mortality associated with the occurrence of a recurrence of VAP in patients hospitalized in the intensive care unit.

An essential first step in this work will be to identify and then use the most consensual definition of recurrence of VAP, encompassing recurrence, persistence and superinfection. We will use the definitions in the protocol for the ASPIC trial, which is currently undergoing enrolment.

The second step is to identify risk factors for recurrence. By identifying these factors, it could be possible to propose a prognostic score that would enable careful monitoring (or modification of antibiotic therapy) of patients most at risk of recurrence. Such a score could then be evaluated in a prospective study.

DETAILED DESCRIPTION:
Ventilator-associated pneumonia (VAP) is a frequent and serious complication in the ICU, defined by the development of a lung infection in patients ventilated for more than 48 hours. The incidence rate of this condition exceeds 18 episodes per 1000 days of mechanical ventilation in Europe. This nosocomial infection is associated with the highest mortality, ranging from 24% to 76% depending on the series. Reducing the incidence of VAP remains a challenge for clinicians, as evidenced by the many recent recommendations that have led to "bundles" to prevent the onset of this complication. Despite this, these recommendations do not propose a strategy to prevent the recurrence of PAVM, a frequent entity with a reported incidence of 25-35% and a non-consensual definition that increases antibiotic consumption, duration of mechanical ventilation and length of stay in the ICU (1,2).

In fact, these recurrences can be linked to:

* Intrinsic patient risk factors (immunosuppression, severity of disease, major inflammatory response, reason for initial admission),
* Inappropriate initial antibiotic therapy (type, duration and dose administered),
* Characteristics specific to the pathogens encountered (virulence factors or resistance),
* Intercurrent complications during management of the initial pneumonia (ARDS, abscess, pleural empyema).

Given the frequency of these recurrences, and the persistent doubts about the role of terrain and pathogen characteristics in their genesis, it seems appropriate to look at risk factors that could help anticipate these events.

The aim of our study will be to identify the risk factors and mortality associated with the occurrence of a recurrence of VAP in patients hospitalized in the intensive care unit.

An essential first step in this work will be to identify and then use the most consensual definition of recurrence of VAP, encompassing recurrence, persistence and superinfection. We will use the definitions in the protocol for the ASPIC trial (3), which is currently undergoing enrolment.

The second step is to identify risk factors for recurrence. By identifying these factors, it could be possible to propose a prognostic score that would enable careful monitoring (or modification of antibiotic therapy) of patients most at risk of recurrence. Such a score could then be evaluated in a prospective study.

1. Combes A, Figliolini C, Trouillet J-L, Kassis N, Dombret M-C, Wolff M, et al. Factors predicting ventilator-associated pneumonia recurrence. Crit Care Med. 2003 Apr;31(4):1102-1107.
2. Combes A, Luyt C-E, Fagon J-Y, Wolff M, Trouillet J-L, Chastre J, et al. Early predictors for infection recurrence and death in patients with ventilator-associated pneumonia. Crit Care Med. 2007 Jan;35(1):146-154.
3. Foucrier A, Roquilly A, Bachelet D, Martin-Loeches I, Bougle A, Timsit JF, Montravers P, Zahar JR, Eloy P, Weiss E; ASPIC study group. Antimicrobial Stewardship for Ventilator Associated Pneumonia in Intensive Care (the ASPIC trial): study protocol for a randomised controlled trial. BMJ Open. 2023 Feb 21;13(2):e065293. doi: 10.1136/bmjopen-2022-065293. PMID: 36810173; PMCID: PMC9944671.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient
* Having presented an episode of ventilator-associated pneumonia defined as the association in a patient undergoing invasive mechanical ventilation ≥ 48h:

  * Radiological signs: two successive chest X-rays showing new or progressive pulmonary infiltrates (in the absence of a medical history of underlying heart or lung disease, a single chest X-ray is sufficient).

    * And at least one of the following signs:
  * Fever > 38.0˚ C without any other cause
  * Leukocytes < 4 × 109 l-1 or > 12 × 109 l-1

    * And at least two of the following signs:
  * Purulent tracheobronchial secretions
  * Cough or dyspnea
  * Decreased oxygenation or increased oxygen requirements, or need for respiratory assistance
* Patient does not object to the use of his/her data for this research

Exclusion Criteria:

* Opposition to the use of personnal data
* People under legal protection (curatorship, guardianship) or safeguard of justice

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults patients having presented an episode of ventilator-associated pneumonia
Sampling Method: Probability Sample
Enrollment: 1569 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-08-31 (Actual); Study Completion 2025-02-26 (Actual)

PRIMARY OUTCOMES:
Mortality at 28 days | 28 days after ICU admission
  Mortality at 28 days, verify if patient died 28 days after Ventilator-associated pneumonia

SECONDARY OUTCOMES:
Number of Ventilator-associated pneumonia recurrences | During inclusion period (from 01JAN2021 to 31DEC2022)
  Number of Ventilator-associated pneumonia recurrences during ICU stay
Number of days without mechanical ventilation at day 28 | 28 days after ICU admission
  Number of days without mechanical ventilation at day 28
Number of days without renal replacement therapy at day 28 | 28 days after ICU admission
  Number of days without renal replacement therapy at day 28
Number of days without catecholamines at day 28 | 28 days after ICU admission
  Number of days without catecholamines at day 28
Number of days without antibiotics at day 28 | 28 days after ICU admission
  Number of days without antibiotics at day 28
MDR acquisition rate | During ICU stay
  multiresistant bacteriaacquisition rate
Length of stay in intensive care unit | During inclusion period (from 01JAN2021 to 31DEC2022)
  Length of stay in intensive care unit
Length of hospital stay | During inclusion period (from 01JAN2021 to 31DEC2022)
  Length of hospital stay
Number of persistent Ventilator-associated pneumonia | During inclusion period (from 01JAN2021 to 31DEC2022)
  Number of persistent Ventilator-associated pneumonia
Number of superinfections of Ventilator-associated pneumonia | During inclusion period (from 01JAN2021 to 31DEC2022)
  Number of superinfections of Ventilator-associated pneumonia

CONTACTS AND LOCATIONS:
Overall Officials: Adrien Bouglé, MD, Study Chair — Hôpital La Pitié-Salpêtrière
Locations (1):
- Hôpital La Pitié-Salpêtrière, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided
unplanned for the moment

REFERENCES:
- [Background] Combes A, Figliolini C, Trouillet JL, Kassis N, Dombret MC, Wolff M, Gibert C, Chastre J. Factors predicting ventilator-associated pneumonia recurrence. Crit Care Med. 2003 Apr;31(4):1102-7. doi: 10.1097/01.CCM.0000059313.31477.2C. PMID 12682479
- [Background] Combes A, Luyt CE, Fagon JY, Wolff M, Trouillet JL, Chastre J. Early predictors for infection recurrence and death in patients with ventilator-associated pneumonia. Crit Care Med. 2007 Jan;35(1):146-54. doi: 10.1097/01.CCM.0000249826.81273.E4. PMID 17080004
- [Background] Foucrier A, Roquilly A, Bachelet D, Martin-Loeches I, Bougle A, Timsit JF, Montravers P, Zahar JR, Eloy P, Weiss E; ASPIC study group. Antimicrobial Stewardship for Ventilator Associated Pneumonia in Intensive Care (the ASPIC trial): study protocol for a randomised controlled trial. BMJ Open. 2023 Feb 21;13(2):e065293. doi: 10.1136/bmjopen-2022-065293. PMID 36810173